CLINICAL TRIAL: NCT02741791
Title: STRIDE-1: A Randomized, Double-blind, Active-controlled Trial to Assess the Efficacy and Safety of AXS-05 Administered Orally to Subjects With Treatment Resistant Major Depressive Disorder
Brief Title: A Study to Assess the Efficacy and Safety of AXS-05 in Subjects With Treatment Resistant Major Depressive Disorder
Acronym: STRIDE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AXS-05-301
Record Dates: First submitted 2016-04-05; First posted 2016-04-18 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Treatment Resistant Major Depressive Disorder
Keywords: AXS-05; Major Depressive Disorder; Treatment Resistant Depression; TRD; MDD; Axsome; NMDA receptor; Refractory depression; Resistant depression; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AXS-05 (Experimental)
  Interventions: Drug: AXS-05
- Bupropion (Active Comparator)
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: AXS-05 — AXS-05 taken daily for 6 weeks.
  Arms: AXS-05
Drug: Bupropion — Buproprion taken daily for 6 weeks.
  Arms: Bupropion

SUMMARY:
To evaluate the efficacy and safety of AXS-05 relative to bupropion in subjects with treatment resistant major depressive disorder (MDD).

This is a randomized, double-blind, active-controlled, 12-week, two-period study consisting of an open-label, bupropion lead-in period, and a double-blind treatment period. The trial is being conducted in subjects with treatment resistant MDD.

Subjects will be considered to have treatment resistant MDD if they have had a historical inadequate response to 1 or 2 antidepressant treatments and a prospective inadequate response to treatment with bupropion during the open-label, lead-in period.

ELIGIBILITY:
Key Inclusion Criteria:

* Currently meets DSM-V criteria for MDD
* History of inadequate response to 1 or 2 adequate antidepressant treatments
* Body mass index (BMI) between 18 and 40 kg/m2, inclusive
* Agree to use adequate method of contraception for the duration of the study
* Additional criteria may apply

Key Exclusion Criteria:

* Suicide risk
* Treatment with any investigational drug within 6 months
* History of electroconvulsive therapy (ECT), vagus nerve stimulation, transcranial magnetic stimulation, or any experimental central nervous system treatment during the current episode or in the past 6 months
* Pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study
* Additional criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2016-03; Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) total score | MADRS change from Baseline to End of Study (6 weeks)
  The MADRS is used to assess depressive symptomatology during the previous week. Subjects are rated on 10 items to assess feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating and lack of interest. Each item is scored on a 7-point scale. A score of 0 indicates the absence of symptoms, and a score of 6 indicates symptoms of maximum severity.

SECONDARY OUTCOMES:
Clinical Global Impressions-Severity (CGI-S) | Baseline to End of Study (6 weeks)
Hamilton Depression Rating Scale - 17 items (HAMD-17) | Baseline to End of Study (6 weeks)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (74):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Beverly Hills, California
  - Garden Grove, California
  - Oakland, California
  - Oceanside, California
  - Panorama City, California
  - Redlands, California
  - Riverside, California
  - San Diego, California
  - San Francisco, California
  - Sherman Oaks, California
  - Temecula, California
  - Upland, California
  - Colorado Springs, Colorado
  - Cromwell, Connecticut
  - Washington D.C., District of Columbia
  - Coral Springs, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Lakeland, Florida
  - North Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Skokie, Illinois
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Nashua, New Hampshire
  - Berlin, New Jersey
  - Cherry Hill, New Jersey
  - Marlton, New Jersey
  - Princeton, New Jersey
  - Toms River, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Jamaica, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Canton, Ohio
  - Dayton, Ohio
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Salem, Oregon
  - Allentown, Pennsylvania
  - Media, Pennsylvania
  - Philadelphia, Pennsylvania
  - Lincoln, Rhode Island
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Wichita Falls, Texas
  - Orem, Utah
  - Charlottesville, Virginia
  - Herndon, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: www.TRDstudy.com — http://www.TRDstudy.com